CLINICAL TRIAL: NCT06900998
Title: A Pilot Study on the Effects of Nimodipine on Alcohol Drinking Among Adults Who Are Heavy Alcohol Drinkers
Brief Title: Effects of Nimodipine on Alcohol Drinking
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000038566; 2P50AA012870-21 (NIH)
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nimodipine (Experimental): All participants will be assigned to this arm and will receive study drug (nimodipine), open label.
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Nimodipine — Nimodipine will be administered orally beginning on the evening prior to the study lab session. 90mg doses will be administered at 6:00pm, 12:00am, 6:00am, and 12:00pm.

SUMMARY:
This is an open label trial aiming to recruit 5 non-treatment seeking adults with Alcohol Use Disorder. All will participate in an alcohol drinking paradigm (ADP) lab session at the Hospital Research Unit (HRU) at Yale-New Haven Hospital (YNHH). Participants will stay overnight and receive nimodipine 90 mg/dose every six hours during an 18-hour period prior to the ADP to allow for the limited central nervous system bioavailability of this drug. Electroencephalogram (EEG) data will be collected before the first dose and after the last dose of nimodipine. Adverse events will be closely monitored during this period. During the ADP session participants will receive a priming dose of alcohol followed by a one-hour monitoring period. This will be followed by three one-hour self-administration periods; during each hour, participants will be able to choose between drinking up to four drinks or receive the monetary equivalents of these drinks (total of 12 drinks over three hours).

DETAILED DESCRIPTION:
This is an open label trial. Five adults, 21-50 years of age, with Alcohol Use Disorder, who are not looking for treatment for their drinking behaviors, and who consume at least 30-70 standard drinks for men or 25-65 standard drinks for women per week will be recruited. Participants will be screened for eligibility including a full physical exam. All will participate in an alcohol drinking paradigm (ADP) lab session at Yale New Haven Hospital's Hospital Research Unit (HRU). Participants will receive nimodipine 90 mg/dose every six hours during an 18-hour period prior to the ADP session while admitted to the HRU overnight. Additionally, electroencephalography (EEG) data will be collected while at the HRU. Nimodipine is rapidly absorbed after oral administration & peak concentrations are achieved within 0.5 to 1.5 hours. However, due to high first-pass metabolism, initial elimination is rapid (equivalent to a half-life of 1-2 hours); consequently, the bioavailability of nimodipine is approximately 13% after oral administration and there is a need for frequent dosing. The terminal elimination half-life of nimodipine is approximately 8 to 9 hours. In order to ensure adequate exposure and CNS bioavailability, the administration schedule used will be similar to that used in the Krupitsky trial. In that study 26 alcohol-dependent patients (who had not consumed alcohol for a month) received treatment with 90 mg dose of nimodipine every 6 hours (4 doses over 18 hours) prior to ketamine administration; results suggest that this dose of nimodipine reduced ketamine-induced psychosis, negative symptoms, euphoria, and sedation as well as the perceived similarity of ketamine effects to alcohol. While the Krupitsky trial did not report any adverse events following exposure to this dose, blood pressure and adverse events will be closely monitored during the treatment period prior to the ADP (monitored at time of each dosing and again 30 minutes, 1 hour, and 2 hours after each dose). During the ADP session, participants will receive a priming dose of alcohol at 1:00pm followed by a one-hour monitoring period. This will be followed by three one-hour self-administration periods; during each hour participants will be able to choose between four drinks or monetary equivalents of these drinks (total of 12 drinks over three hours).

After the ADP, participants will be given dinner, and breath alcohol levels will be assessed until 10pm. If at 10pm, a participant has a breath alcohol level less than .03, they will be discharged; if greater than .03 but less than .05, a nurse on the clinical unit will evaluate to ensure the participant is alert and oriented and has no visible signs of intoxication (slurred speech, unsteady gait). If cleared by the nurse, instructions will be given to not drive or operate heavy machinery for the rest of the night. If not cleared, the nurse will continue to monitor until clearance is given. All participants will then be discharged and provided an Uber ride home.

Participants will have 2 follow-up visits 1-week and 1-month after the ADP session.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-50 (The lower limit is to avoid offering alcohol to individuals below the drinking age of 21. The upper age is determined by experience recruiting for our prior studies).
2. Ability to read English at 6th grade level or higher.
3. Meet DSM-V criteria for at least moderate AUD.
4. Average weekly alcohol consumption of 30-70 standard drinks for men and 20-65 drinks for women. The lower limits are consistent with the lower sex-specific cut-offs defining high-risk drinking based on World Health Organization Risk Levels (WHO, 2000); the upper limits are designed to avoid recruiting participants whose drinking is likely to exceed the number of drinks available in the alcohol drinking paradigm (ADP).

Exclusion Criteria:

1. Individuals who are seeking alcohol treatment or have been in alcohol treatment within the past 6 months.
2. Meet current DSM-V criteria for substance use disorder, except for tobacco use disorder or mild cannabis use disorder.
3. Positive urine drug screens at more than 1 baseline appointment for opiates, cocaine, benzodiazepines, and barbiturates.
4. Psychotic or other severe psychiatric disorders as determined by clinical evaluation.
5. Regular use of psychoactive drugs, except for individuals on a stable dose of an antidepressant for at least 2 months.
6. Medical conditions that would contraindicate the consumption of alcohol or use of nimodipine including untreated or not adequately controlled hypertension or hypotension. Blood pressure at or below 100/65 will be exclusionary.
7. Clinically significant abnormalities in screening laboratories, including aspartate aminotransferase (AST) >3 times upper limit of normal (ULN); alanine aminotransferase (ALT) > 3 times ULN; total bilirubin >1.5 times ULN; serum creatinine >2.0 times ULN.
8. Concurrent use of the following medications: CYP3A4 inhibitors and inducers, other calcium channel blockers, or other blood pressure lowering medications.
9. Neurological trauma or disease, delirium, or hallucinations, or clinically significant or unstable medical conditions, including uncontrolled hypertension or diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic diseases, which in the opinion of the study physician and PI, may put the patient at risk because of participation in the study.
10. Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) scores of 8 or greater or a history of significant repeated alcohol withdrawals to reduce the likelihood of withdrawal symptomatology if subjects reduce their drinking.
11. Women who are pregnant or nursing.
12. Participants who refuse to use a reliable method of birth control from the time of first medication administration to 7 days after. These include oral contraceptives, contraceptive sponge, patch, double barrier (diaphragm/spermicidal or condom/spermicidal), intrauterine contraceptive system, etonogestrel implant, medroxyprogesterone acetate contraceptive injection, complete abstinence from sexual intercourse, hormonal vaginal contraceptive ring, surgical sterilization, or true abstinence.
13. Subjects who report disliking spirits will be excluded because hard liquor will be provided during the ADP.
14. Subjects who have taken any investigational drug within 4 weeks of the anticipated date of the first study dose.
15. Individuals who report heavy drinking days in the 2 days prior to their intake appointment but have a negative ethyl glucuronide (EtG) test to rule out subjects who are misrepresenting their drinking history.
16. Subjects who have donated blood within the past 6 weeks.
17. Heart rate of less than 50 bpm.
18. Subjects with a history or presence of cirrhosis.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of drinks consumed | Lab Session 1 (Day 1)
  Total number of drinks (out of 12) that were consumed during the alcohol drinking paradigm (ADP) session.
Alcohol Craving using Yale Craving Scale | Lab Session 1 (Day 1)
  Craving for alcohol based on Yale Craving Scale, scores ranging from 0-112 mm on a visual analog scale, with higher measurements indicating higher craving.
Stimulation Effect | Lab Session 1 (Day 1)
  Stimulation effect collected using the Biphasic Alcohol Effect Scale. Brief Biphasic Alcohol Effects Scale-Stimulation subscale, measuring stimulation effects of alcohol on an 11-point rating scale from 0=Not at All to 10=Extremely, total scores ranging from 0 - 30, with higher measurements indicating higher stimulation.
Sedation Effect | Lab Session 1 (Day 1)
  Stimulation effect collected using the Biphasic Alcohol Effect Scale. Brief Biphasic Alcohol Effects Scale-Sedation subscale, measuring sedation effects of alcohol on Day 7, 6 items, 11-point rating scale from 0=Not at All to 10=Extremely, total scores ranging from 0 - 30, with higher measurements indicating higher sedation.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Lab Session 1 (Days 0 and 1)
  Mean change in systolic blood pressure in mmHg
Change in Diastolic Blood Pressure | Lab Session 1 (Days 0 and 1)
  Mean change in diatolic blood pressure in mmHg
Change in Heart Rate | Lab Session 1 (Days 0 and 1)
  Mean change in heart rate measured in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Principal Investigator — Yale University School of Medicine, Dept of Psychiatry
Locations (1):
- Yale University School of Medicine (Connecticut Mental Health Center), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study done to inform procedures for a larger clinical trial. There are no plans to share IPD at this time.

REFERENCES:
- [Background] Krupitsky EM, Burakov AM, Romanova TN, Grinenko NI, Grinenko AY, Fletcher J, Petrakis IL, Krystal JH. Attenuation of ketamine effects by nimodipine pretreatment in recovering ethanol dependent men: psychopharmacologic implications of the interaction of NMDA and L-type calcium channel antagonists. Neuropsychopharmacology. 2001 Dec;25(6):936-47. doi: 10.1016/S0893-133X(01)00346-3. PMID 11750186